CLINICAL TRIAL: NCT02569515
Title: An Open-Label Study of the Tolerability and Flexibility of Multi-Dose NeoRecormon Administered by Reco-Pen in Pre-Dialysis Patients With Chronic Renal Anemia.
Brief Title: A Study of Epoetin Beta (NeoRecormon) in Predialysis Patients With Renal Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18101
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (1):
- Epoetin Beta (Experimental): Patients will be administered 3 times (X) 30 International unis per kilogram(IU/Kg body weight per week of eopetin beta subcurtaneously using the device RecoPen. The dosage could be increased every 4 weeks by 3 X20 IU/Kg.
  Interventions: Drug: Epoetin Beta

INTERVENTIONS:
Drug: Epoetin Beta — Initial dose: 3X30 IU/Kg body weight administered subcutaneously using RecoPen. Dosage could be increased by 3X20 IU/Kg every 4 weeks up to a maximum of 720 IU/Kg per week.
  Other Names: NeoRecormon

SUMMARY:
This study will evaluate the tolerability, and effect on quality of life, in patients receiving multi-dose NeoRecormon administered by RecoPen in predialysis patients with chronic renal anemia. The anticipated time on study treatment is 10 months, and the target sample size is 60 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-65 years of age
* Chronic renal failure (Stages I-III)
* No previous epoetin therapy

Exclusion Criteria:

* Poorly controlled hypertension
* History or evidence of malignancy
* Relevant acute or chronic bleeding (requiring therapy) within 3 months before study drug
* Women who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participantss who change to once weekly NeoRocormon | 10 months
Percentage of participants with local intolerabilities (pain/allergic reactions) | 10 months
Percentage of participants who withdrew due to inability to use RecoPen | 10 months
Percentage of participants who changed dose during treatmnent | 10 months

SECONDARY OUTCOMES:
Quality of life evaluated by the Short Form 36 | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (2):
- Bulgaria (2):
  - Sofia
  - Varna